CLINICAL TRIAL: NCT07178262
Title: Opioid Sparing Effect of Erector Spinae Block in Patients Undergoing Total Abdominal Hysterectomy; A Randomized Control Trial
Brief Title: Erector Spinae Block in Reducing Peri-operative Opioid Consumption in Total Abdominal Hystrectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kulsoom International Hospital (Other)
Responsible Party: Principal Investigator, Waqas Anjum, Principal Investigator, Kulsoom International Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERC-030
Record Dates: First submitted 2025-08-31; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Erector Spinae Block; Enhanced Recovery After Surgery (ERAS) Protocol; Opioid
MeSH Terms: interventions — Parapsychology; Dental Occlusion; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Erector spinae group (Active Comparator): Patients in this group will receive bilateral erector spinae block at T10 level using 30ml of 0.25% Bupivacaine before surgical incision.
  Interventions: Drug: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®)
- Placebo (Placebo Comparator): Patient in this group will receive Norma saline in Erector spinae block at T10 level bilaterally before surgical incision.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®) — Bilateral Erector Spinae Block at T10 level using 30ml of 0.25% Bupivacaine will be administered under Ultrasound guidance before surgical incision.
  Arms: Erector spinae group
Drug: Placebo — Bilateral Erector Spinae Block at T10 level using 30ml of Normal saline will be administered under Ultrasound guidance before surgical incision.
  Arms: Placebo

SUMMARY:
Hystrectomy is a surgical procedure that involves removal of uterus from the body of patient using a lower abdominal incision. This is an extremely painful procedure which causes discomfort and greatly increases opioids consumption in the peri-operative period. This can be reduced by using nerve blocks such as Erector spinae plane block.

DETAILED DESCRIPTION:
Total abdominal hystrectomy is associated with significant pain due to large abdominal incision and significant surgical dissection. This greatly increases the consumption of Opioid in the peri-operative period. High dose opioid consumption is associated with constipation, nausea, vomiting and respiratory depression. This significantly hampers post operative recovery. Fascial plane blocks such as Erector spinae block provides significant analgesia greatly reducing opioid consumption and there by reducing the associated side effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class: I, II and III .
* Elective Hysterectomy under General Anesthesia.

Exclusion Criteria:

* Lack of consent
* Body mass index >35 kg/m2
* Allergic to study medicine
* Opioid abuse or misuse disorder
* Chronic pain

Ages: 16 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Total Intra-operative Fentanyl consumption | From surgical incision till end of surgery

SECONDARY OUTCOMES:
Total amount of IV Tramadol consumed in post operative period | First 24 hours after surgery
Post operative pain score | Baseline that is pain score upon arrival in post anesthesia care unit in the post operative period and then at 1hours ,2 hours ,4 hours,6 hours,12 hours and 24 hours in the post operative period
  This will be assessed Visual Analog Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Kulsoom Internation Hospital, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamed MA, Boules ML, Mahmoud MAEM, Abdelghaffar RA. The effect of erector spinae plane block on fentanyl consumption during open abdominal hysterectomy: a randomised controlled study. BMC Anesthesiol. 2023 Jun 5;23(1):194. doi: 10.1186/s12871-023-02156-3. PMID 37277703